CLINICAL TRIAL: NCT03406442
Title: Endoscopic Endonasal Transpterygoid Approaches
Brief Title: Transpterygoid Approaches
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed El-Rahman Mohamed Azzam, Dr.Ahmed EL-rahman Mohamed Azzam, Assistant lecture of otorhinolaryngology department, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: transpterygoid approaches
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Transpterygoid Approaches

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients (Other): The patient who have lesions affecting pterygopalatine fossa, lateral recess of the sphenoid sinus, petrous apex, Meckel's cave, cavernous sinus, infratemporal fossa and lateral nasopharynx and can be treated by endonasal endoscopic transptergoid approaches
  Interventions: Procedure: Transpterygoid approaches

INTERVENTIONS:
Procedure: Transpterygoid approaches — All patients will be operated by transpterygoid approaches which is classified into 5 major types.Type A involves thinning of the pterygoid process to access to Pterygopalatine fossa. Type B involves the removal of the medial and anterior aspect of the base of the pterygoid process to access the lateral recess of sphenoid sinus. Type C involves removing the base of the pterygoid plates to reach the petrous apex, Meckel's cave, or cavernous sinus. Type D requires removal of the pterygoid plates to access the infratemporal fossa. Type E requires the removal of the medial pterygoid plate or the entire pterygoid process, and the medial third of the Eustachian tube to acessof the lateral nasopharynx

SUMMARY:
To identify:

1. The most frequent pathologies affecting pterygopalatine fossa, lateral recess of the sphenoid sinus, petrous apex, Meckel's cave, cavernous sinus, infratemporal fossa and lateral nasopharynx that can be treated by endonasal endoscopic transptergoid approaches, the most common presenting manifestations and indication of surgery.
2. The different techniques and feasibility of different endonasal endoscopic transpterygoid approaches and the frequency of utilization of approach.
3. Try to establish a protocol for post-operative care and management of complications.
4. Obtain sufficient surgical experience in endonasal endoscopic transpterygoid surgery to establish endonasal endoscopic skull-base surgery in Assiut University Hospital.

DETAILED DESCRIPTION:
Skull base surgery has undergone dramatic advances. During early stages, the endoscopic approaches were limited by the resultant skull base defects .

Access to the pterygopalatine fossa (PPF) is a surgical challenge due to its deep location in the mid-third of the face and its complex array of vascular and neural structures. An important aspect of the PPF is its topographical relation to the orbit and cranial cavity.

The philosophy behind the transpterygoid approach centers on the maxillary sinus as the primary corridor, displaces the contents of the PPF and removes the pterygoid process partially or completely to reach to the lateral extent of the endonasal technique.

The endoscopic endonasal transpterygoid approaches classified into five types. Type A involves thinning of the pterygoid process to gain access to PPF. Type B involves removal of the medial and anterior aspect of the base of the pterygoid process to access the lateral recess of the sphenoid sinus. Type C involves dissecting the vidian nerve to identify the petrous ICA and removing the base of the pterygoid plates to reach the petrous apex, Meckel's cave, or cavernous sinus. Type D requires a variable removal of the pterygoid plates to access the infratemporal fossa. Type E requires removal of part or even the entire pterygoid process, and the medial third of the Eustachian tube to provide exposure of the lateral nasopharynx.

ELIGIBILITY:
Inclusion Criteria:

Any patient with lesions affecting pterygopalatine fossa, lateral recess of the sphenoid sinus, petrous apex, Meckel's cave, cavernous sinus, infratemporal fossa and lateral nasopharynx that can be treated by endonasal endoscopic transptergoid approaches.

Exclusion Criteria:

1. Medically unfit patients for surgery
2. In case of distant metastasis in tumors

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Type of the pathology | 1 week
  Identification of the type lesion will be made.
Frequency of residual mass | 1 week
  Early MRI will be obtained after a week to asses the extent of resection and search if there is residual mass.
Frequency of recurrence | 6 months
  Imaging will be done in six months period to search for any recurrence.
Frequency of complication | 1 month
  Post-operative follow up of the patients will be done to identify the frequency of complication either rhinogenic as bleeding , synechiae, csf leakage or orbital complication as proptosis, visual affection or intracranial complication as meningitis.
Operation time | intraoperative
  The time of the operation will be calculated in this endoscopic approach comparing to traditional open technique.
Intraoperative bleeding | Intraoperative
  The amount of intraoperative bleeding and the ability to control it.
Surgical field exposure | Intraoperative
  The possibility of the approach to reach lesions affecting deep area in the skull as pterygopalatine fossa, lateral recess of the sphenoid sinus, petrous apex, Meckel's cave, cavernous sinus, infratemporal fossa and lateral nasopharynx.
Post-operative stay | 2 weeks
  post-operative stay of the patient in hospital.
mortality rate | 1 year
  any deaths

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Shaker Abd-Elaal, MD, Study Chair — Assiut University; Hossam El-din Mahmoud El-Bosraty, MD, Principal Investigator — Cairo University; Mohamed Modather Abd El-Naam, MD, PHD, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chibbaro S, Cornelius JF, Froelich S, Tigan L, Kehrli P, Debry C, Romano A, Herman P, George B, Bresson D. Endoscopic endonasal approach in the management of skull base chordomas--clinical experience on a large series, technique, outcome, and pitfalls. Neurosurg Rev. 2014 Apr;37(2):217-24; discussion 224-5. doi: 10.1007/s10143-013-0503-9. Epub 2013 Nov 19. PMID 24249430
- [Background] Choi J, Park HS. The clinical anatomy of the maxillary artery in the pterygopalatine fossa. J Oral Maxillofac Surg. 2003 Jan;61(1):72-8. doi: 10.1053/joms.2003.50012. PMID 12524612
- [Background] Kasemsiri P, Solares CA, Carrau RL, Prosser JD, Prevedello DM, Otto BA, Old M, Kassam AB. Endoscopic endonasal transpterygoid approaches: anatomical landmarks for planning the surgical corridor. Laryngoscope. 2013 Apr;123(4):811-5. doi: 10.1002/lary.23697. PMID 23529878
- [Background] Hofstetter CP, Singh A, Anand VK, Kacker A, Schwartz TH. The endoscopic, endonasal, transmaxillary transpterygoid approach to the pterygopalatine fossa, infratemporal fossa, petrous apex, and the Meckel cave. J Neurosurg. 2010 Nov;113(5):967-74. doi: 10.3171/2009.10.JNS09157. Epub 2009 Nov 20. PMID 19929194
- [Background] Kassam AB, Prevedello DM, Carrau RL, Snyderman CH, Thomas A, Gardner P, Zanation A, Duz B, Stefko ST, Byers K, Horowitz MB. Endoscopic endonasal skull base surgery: analysis of complications in the authors' initial 800 patients. J Neurosurg. 2011 Jun;114(6):1544-68. doi: 10.3171/2010.10.JNS09406. Epub 2010 Dec 17. PMID 21166570